CLINICAL TRIAL: NCT06309407
Title: Dosimeter Location and Measured Effective Radiation Dose in Pain Management Physicians
Brief Title: Dosimeter Location in Pain Physicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Sandy Christiansen, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00024903
Record Dates: First submitted 2024-02-22; First posted 2024-03-13 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: RAD
Keywords: Dosimeter; Radiation; Pain Medicine; Physician

STUDY DESIGN:
Intervention Model Description: Participants were randomized to wear either chest dosimeters only or chest and hand dosimeters for the duration of the study in order to measure differences in radiation readings by each dosimeter location.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Chest and Hand Dosimeters (Experimental): Subjects will wear both chest and hand dosimeters during all radiation procedures performed at the Comprehensive Pain Center during the study period.
  Interventions: Device: Hand Dosimeters
- Chest Dosimeter (Active Comparator): Subjects will wear only a chest dosimeter during all radiation procedures performed at the Comprehensive Pain Center during the study period.
  Interventions: Device: Standard Practice

INTERVENTIONS:
Device: Hand Dosimeters — Participants were assigned to wear hand dosimeters in addition to the standard chest dosimeter worn by all participants
  Arms: Chest and Hand Dosimeters
Device: Standard Practice — Participants only wore standard chest dosimeters
  Arms: Chest Dosimeter

SUMMARY:
The primary objective is to determine if there is a significant difference in radiation readings between dosimeters worn on the chest versus the hand of interventional pain management physicians and elucidate which dosimeter had higher readings.

The secondary objective is to track incidences of physician glove breaches in both groups to assess if wearing hand dosimeters is associated with an increased risk of this event.

ELIGIBILITY:
Inclusion Criteria:

* Physicians actively performing fluoroscopy procedures at the Comprehensive Pain Center.

Exclusion Criteria:

* Those that do not want to participate in the quality improvement project.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Christiansen, MD, Principal Investigator — Associate Professor
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared with other researchers.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants were randomized. There were no participants excluded before assignment to groups.
Period: Overall Study
Arm/Group | Chest and Hand Dosimeters | Chest Dosimeter
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chest and Hand Dosimeters | Chest Dosimeter | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 4 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Radiation Readings
Description: Dose equivalent in mREM for each dosimeter that is worn by the subject.
Time Frame: 6 months
Population: In the chest and hand dosimeter group, for each participant one chest and one hand dosimeter recording was analyzed. In the chest group, one chest dosimeter recordings was analyzed.
Measure: Mean (95% Confidence Interval); unit: mREM
Units Other Than Participants: Dosimeters
Arm/Group | Chest and Hand Dosimeters | Chest Dosimeter
Number analyzed (Participants) | 5 | 5
Number analyzed (Dosimeters) | 10 | 5
mREM
  Chest Dosimeters: number analyzed (Dosimeters) | 5 | 5
  Chest Dosimeters | 122.8 [62.4 to 183.2] | 158.8 [40.5 to 277.1]
  Hand Dosimeters: number analyzed (Participants) | 5 | 0
  Hand Dosimeters: number analyzed (Dosimeters) | 5 | 0
  Hand Dosimeters | 236.9 [80.7 to 393.3] |

2. Secondary Outcome: Total Number of Glove Breach Events
Description: Number of intra-procedure glove breaches
Time Frame: 6 months
Measure: Number; unit: Number of Glove Breach Events
Arm/Group | Chest and Hand Dosimeters | Chest Dosimeter
Number analyzed (Participants) | 5 | 5
Number of Glove Breach Events | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Chest and Hand Dosimeters | Chest Dosimeter
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Small sample size that is not powered to detect a difference.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT06309407/Prot_SAP_000.pdf